CLINICAL TRIAL: NCT01721304
Title: Decision Making Among Treatment Alternatives for Abnormal Uterine Bleeding (AUB)
Brief Title: Decisionmaking for Abnormal Uterine Bleeding (AUB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lisa Hess, Assistant Professor of Medicine and Public Health, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1009001853 (0904-66B)
Record Dates: First submitted 2012-10-25; First posted 2012-11-05 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Abnormal Uterine Bleeding
Keywords: decision making; abnormal uterine bleeding; adaptive conjoint analysis; satisfaction; regret
MeSH Terms: conditions — Metrorrhagia; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive Conjoint Analysis (Experimental): Computerized survey to elicit preferences
  Interventions: Other: Adaptive Conjoint Analysis
- Usual care (No Intervention): Patients are counseled by their physician as usual

INTERVENTIONS:
Other: Adaptive Conjoint Analysis — Computerized survey to elicit patient preferences
  Arms: Adaptive Conjoint Analysis

SUMMARY:
The purpose of this study is to determine if using a computer survey about preferences for treatment of abnormal uterine bleeding (AUB) is useful and if it will improve patient satisfaction with clinical care and decision making. This study is a two-part study. The first pilot tests the computerized tool to ensure it is understood by patients, then the second part is a randomized study (computerized tool versus usual care) to see if improvements are made in satisfaction and if there are reductions in decision regret.

DETAILED DESCRIPTION:
The purpose of this study is to determine if using a computer survey about preferences for treatment of abnormal uterine bleeding (AUB) is useful and if it will improve patient satisfaction with clinical care and decision making. This study was designed to develop and test the use of ACA as part of routine clinical care for women diagnosed with AUB. After pilot testing, the ACA survey is administered in this study where patients are assigned to receive the ACA or to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of dysfunctional or abnormal uterine bleeding (AUB) that is recommended for treatment
* Have not yet selected or initiated treatment for current AUB diagnosis
* Be at least 18 years of age.
* Be possible candidates for either medical or surgical therapy
* Able to provide informed consent for treatment options for oneself

Exclusion Criteria:

* Are currently being treated for cancer
* Any cancer diagnosis within the past 2 years (other than non-melanoma skin cancer)
* AUB due to serious pelvic pathology, medications, pregnancy or systemic disease that limits their range of treatment options
* Are not recommended for surgical intervention
* Are not recommended for medical intervention
* Are under 18 years of age
* Have not received a diagnosis of AUB
* Are currently being treated for AUB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Differences in patient-reported satisfaction between treatment groups | 6 weeks
  Satisfaction with care as measured by the Functional Assessment of Chronic Illness Therapy-Treatment Satisfaction-Patient Scale (FACT-TS-PS)
Differences in decision regret between treatment groups | 6 weeks
  Decision regret is measured by the Decision Regret Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Hess, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Southern Pines Women's Health Center, Southern Pines, North Carolina

REFERENCES:
- [Result] Hess LM, Litwiller A, Byron J, Stutsman J, Kasper K, Learman LA. Preference elicitation tool for abnormal uterine bleeding treatment: a randomized controlled trial. Patient. 2015 Apr;8(2):217-27. doi: 10.1007/s40271-014-0078-8. PMID 25074354
- See also: Preference elicitation tool for abnormal uterine bleeding treatment: a randomized controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/25074354